CLINICAL TRIAL: NCT01298726
Title: Pharmaceutical Care Program for Users of Brazilian Public Health Care System With Type 2 Diabetes Mellitus: Randomized Controlled Clinical Trial
Brief Title: Pharmaceutical Care in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Ouro Preto (Other)
Responsible Party: LISIANE DA SILVEIRA EV, UNIVERSIDADE FEDERAL DE OURO PRETO
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0040.0.238.000-09
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-01

CONDITIONS: DIABETES MELLITUS, TYPE 2
Keywords: PHARMACEUTICAL SERVICES; DIABETES MELLITUS
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PHARMACEUTICAL CARE (Other)
  Interventions: Other: PHARMACEUTICAL CARE
- HEALTH USUAL CARE (Other)
  Interventions: Other: HEALTH USUAL CARE

INTERVENTIONS:
Other: PHARMACEUTICAL CARE — The pharmaceutical care program was characterized by face to face monthly visits to collect information, register information, prepare plan of care for every health problem; identification of drug therapy problems, communication to prescribers the drug therapy problems identified and education of participants to resolve the drug therapy problems.
  Arms: PHARMACEUTICAL CARE
Other: HEALTH USUAL CARE — Usual care as defined in health consultations with doctors, nutritionists and nurses, access to laboratory tests and essential medicines
  Arms: HEALTH USUAL CARE

SUMMARY:
The purpose of this study is to examine the effect of a pharmaceutical care program on the level of glycated hemoglobin for hyperglycemic users of brazilian public health care system in drug treatment for type 2 diabetes.

DETAILED DESCRIPTION:
The chronic diseases, including diabetes mellitus (DM) are a major public health problems of today. There is evidence that glycated hemoglobin (A1C) levels above 7% are associated with a progressively greater risk of chronic complications related to DM. However, approximately 60% of diabetics do not achieve glycemic control. In Brazil, pharmacists are not involved in direct care of patients with DM. The investigators conducted a randomized controlled trial, for six months, in Ouro Preto, Minas terais to determine the effect of pharmaceutical intervention on glycemic control in patients with diabetes and hyperglycemic (A1C > 7%). One hundred and twenty-nine subjects were randomized to receive usual care only or usual care and pharmaceutical intervention. The population of those who had access in the brazilian public health care system, as consultations with doctors, nurses and nutritionists, laboratory tests and access to essential medicines were considered as conventional health care.

ELIGIBILITY:
Inclusion Criteria:

* MINIMAL AGE 18 YEARS OLD
* USE OF DIABETES ORAL MEDICATION
* MINIMAL GLYCOHEMOGLOBIN 7%

Exclusion Criteria:

* PREGNANT AND NURSING WOMEN
* PEOPLE UNABLE TO ATTEND THE STUDY SITE
* PARTICIPANTS OF OTHER PROGRAMS OF PHARMACEUTICAL CARE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
GLYCATED HEMOGLOBIN (A1C) LEVELS | AT THE BEGINNING AND END OF STUDY (AFTER 6 MONTHS OF THE START)
  glycated hemoglobin levels was determined in the laboratory by high-performance liquid chromatography (HPLC) using venous blood as a sample

SECONDARY OUTCOMES:
FASTING GLUCOSE LEVELS | AT THE BEGINNING AND END OF STUDY (AFTER 6 MONTHS OF THE START)
  fasting glucose levels was determined in the laboratory by enzymatic colorimetric method using venous blood as a sample
TOTAL CHOLESTEROL LEVELS | AT THE BEGINNING AND END OF STUDY (AFTER 6 MONTHS OF THE START)
  total cholesterol levels was determined in the laboratory by enzymatic colorimetric method using venous blood as a sample
LDL CHOLESTEROL LEVELS | AT THE BEGINNING AND END OF STUDY (AFTER 6 MONTHS OF THE START)
  LDL levels was determined in the laboratory by enzymatic colorimetric method using venous blood as a sample
HDL CHOLESTEROL LEVELS | AT THE BEGINNING AND END OF STUDY (AFTER 6 MONTHS OF THE START)
  HDL levels was determined in the laboratory by enzymatic colorimetric method using venous blood as a sample
TRIGLYCERIDES LEVELS | AT THE BEGINNING AND END OF STUDY (AFTER 6 MONTHS OF THE START)
  triglycerides levels was determined in the laboratory by enzymatic colorimetric method using venous blood as a sample
SYSTOLIC BLOOD PRESSURE LEVELS | AT THE BEGINNING AND END OF STUDY (AFTER 6 MONTHS OF THE START)
  blood pressure levels was determined by indirect method with digital sphygmomanometer, Omron HEM 742
DIASTOLIC BLOOD PRESSURE LEVELS | AT THE BEGINNING AND END OF STUDY (AFTER 6 MONTHS OF THE START)
  blood pressure levels was determined by indirect method with digital sphygmomanometer, Omron HEM 742

CONTACTS AND LOCATIONS:
Overall Officials: LISIANE S EV, DR, Study Chair — Universidade Federal de Ouro Preto; ANDREA G GRABE, DR, Study Director — Universidade Federal de Ouro Preto
Locations (1):
- Universidade Federal de Ouro Preto, Ouro Preto, Minas Gerais, Brazil